CLINICAL TRIAL: NCT03488121
Title: When Less is More: A Real World Randomized Controlled Study to Incentivize Doctors for Appropriate Use of Medical Care in NL
Brief Title: Randomized Controlled Study to Incentivize Doctors for Appropriate Use of Medical Care in NL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to logistical reasons
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Hai Van Nguyen, Assistant Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017.282
Record Dates: First submitted 2018-03-28; First posted 2018-04-04 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2018-09

CONDITIONS: Prescription Practices of Family Physicians in NL

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Poster Only (Experimental): This arm will only receive motivational posters.
  Interventions: Behavioral: Poster
- Thank-you Letter Only (Experimental): This arm will only receive thank-you letters.
  Interventions: Behavioral: Thank-you Letter
- Double Incentive (Experimental): This arm will receive both motivational posters and thank-you letters.
  Interventions: Behavioral: Poster; Behavioral: Thank-you Letter
- Control (No Intervention): This arm will not receive any intervention.

INTERVENTIONS:
Behavioral: Poster — Posters contain inspirational messages and pictures highlighting the important and unique roles that patients and physicians can play in reducing unnecessary care and health care costs. These posters will be placed in physician offices.
  Arms: Double Incentive; Poster Only
Behavioral: Thank-you Letter — Physicians will be sent thank-you letters containing changes in the rates of antibiotics and serum ferritin tests ordered since introduction of Choosing Wisely NL and a thank-you message from the NL Medical Association.
  Arms: Double Incentive; Thank-you Letter Only

SUMMARY:
Choosing Wisely Canada is a campaign for promoting appropriate use of medical services to reduce unnecessary prescribing and unnecessary diagnostic tests. Its success depends on physicians' uptake of the campaign's recommendations on appropriate use of health care. This study will conduct a cluster-randomized controlled trial to evaluate the effects of two low-cost incentives for physicians to promote their uptake of Choosing Wisely recommendations in Newfoundland and Labrador (NL). The first incentive involves placing a motivational poster in a physician's examination room. These posters will contain motivational messages about the important roles that doctors and patients can play in reducing unnecessary care. The second incentive involves sending thank-you letters to physicians to recognize their contribution in reducing unnecessary care, and thus, 'nudge' them into following recommendations. The study will evaluate the effects of the incentives on physicians' prescribing of antibiotics and serum ferritin tests. Potential cost savings of implementing the two incentives will also be estimated.

DETAILED DESCRIPTION:
The study will employ a prospective, cluster randomized controlled trial design and will involve fee-for-service family physicians in NL. Randomization will be performed at the clinic level and stratified by clinic size. Clinics will be randomized into one of four groups: i) the control group will not receive any incentive; ii) the poster group will receive posters only; iii) the letter group will receive thank-you letters only; and iv) the double incentive group will receive both posters and thank-you letters. The number of clinics in each group will be equal.

The study will test two interventions. First, it will examine the impact of placing a poster in a physician's examination room containing motivational messages about the important roles that doctors and patients can play in reducing unnecessary care. The second incentive will involve sending thank-you letters to physicians aiming to encourage them to following Choosing Wisely's recommendations by recognizing their contribution in reducing unnecessary care. The study will focus on physicians' prescribing of antibiotics and serum ferritin tests. The posters will be designed to contain inspirational messages and pictures that highlight the important and unique roles that physicians and patients play in reducing unnecessary care and health care costs. These will be displayed in physicians' examination rooms so that they are salient to doctors and patients. The thank-you letters will contain two types of information: the changes in the rates of antibiotics and serum ferritin tests ordered since Choosing Wisely NL's introduction and a thank you message from the NL Medical Association (NLMA). These will be sent to doctors quarterly (to reinforce the message) with the changes in the rates of antibiotics and serum ferritin tests ordered being updated.

These incentives will be delivered over a 12-month period. The researchers will measure changes in the study outcomes at the end of this 12-month intervention period. Further, to examine if the effects of the intervention are sustained, these changes will be evaluated again 6 months after the withdrawal of incentives. The two incentives will be delivered via NLMA to its member family physicians. As such, physicians will be blinded to this study (i.e., they would not know that these posters and letters are part of a study). The study will focus on fee-for-service physicians in NL as data on the number of patients are only available for these physicians.

ELIGIBILITY:
Inclusion Criteria:

* All Fee-For-Service family physicians registered with the NL Medical Association

Exclusion Criteria:

* Salary based family physicians

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of antibiotic prescriptions | 12 months
  Rate of antibiotic prescriptions will be calculated as the number of antibiotic prescriptions per patient.
Rate of ordering of serum ferritin tests | 12 months
  Rate of serum ferritin tests ordered will be calculated as the number of serum ferritin tests ordered per patient.

SECONDARY OUTCOMES:
Cost savings from implementing the incentives | 12 months
  Cost savings for 'Poster Only' arm: To estimate cost savings for this arm, reductions in prescription of antibiotics and serum ferritin tests in this arm (relative to control arm) estimated by the RCT will be converted into monetary values using pricing data from the literature.
  Cost savings for 'Thank-you Letter Only' arm: To estimate cost savings for this arm, reductions in prescription of antibiotics and serum ferritin tests in this arm (relative to control arm) estimated by the RCT will be converted into monetary values using pricing data from the literature.
  Cost savings for 'Double Incentive' arm: To estimate cost savings for this arm, reductions in prescription of antibiotics and serum ferritin tests in this arm (relative to control arm) estimated by the RCT will be converted into monetary values using pricing data from the literature.
  Total cost savings will then be compared with total cost of implementing the associated incentive to estimate total net cost savings.

CONTACTS AND LOCATIONS:
Overall Officials: Hai Nguyen, PhD, Principal Investigator — Memorial University of Newfoundland
Locations (1):
- School of Pharmacy, Memorial University of Newfoundland, St. John's, Newfoundland and Labrador, Canada